CLINICAL TRIAL: NCT03971227
Title: Clinical Evaluation of Safety and Effectiveness for the Acuity 200 (Fluoroxyfocon A) Rigid Gas Permeable Contact Lens
Brief Title: Clinical Evaluation of Acuity 200 (Fluoroxyfocon A) RGP Contact Lens
Acronym: Acuity 200
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Acuity Polymers, Inc. (Industry)
Collaborators: Andre Vision and Device Research (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AVDR 2019-02 v1.0
Record Dates: First submitted 2019-05-30; First posted 2019-06-03 (Actual); Last update posted 2020-05-12 (Actual); Status verified 2020-01

CONDITIONS: Refractive Errors
Keywords: refractive; permeable; lens; rigid; gas; myopia
MeSH Terms: conditions — Refractive Errors; Muscle Rigidity; Mucopolysaccharidosis IV; Myopia | interventions — Contact Lenses

STUDY DESIGN:
Intervention Model Description: This is an open-label, multi-center, randomized concurrent-control study with the treatment duration of 90 days.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Acuity 200 contact lens (Experimental): Rigid gas permeable contact lens for daily wear, fluoroxyfocon A
  Interventions: Device: Acuity 200 (Fluoroxyfocon A) contact lens
- Acuity 100 contact lens (Active Comparator): Rigid gas permeable contact lens for daily wear, hexafocon A
  Interventions: Device: Acuity 100 (Hexafocon A) contact lens

INTERVENTIONS:
Device: Acuity 200 (Fluoroxyfocon A) contact lens — Daily wear rigid gas permeable contact lens
  Arms: Acuity 200 contact lens
Device: Acuity 100 (Hexafocon A) contact lens — Daily wear rigid gas permeable contact lens
  Arms: Acuity 100 contact lens

SUMMARY:
The objective of this clinical investigation is to collect valid scientific safety and effectiveness data on the Acuity 200 (fluoroxyfocon A) Rigid Gas Permeable Contact Lens, manufactured from a newly developed rigid gas permeable material that is highly permeable to oxygen. The clinical performance data reported from this study is intended to be submitted to the U.S. Food and Drug Administration Center for Devices and Radiological Health (CDRH) in support of a 510(k) premarket notification.

DETAILED DESCRIPTION:
This is an open-label, multi-center, randomized concurrent-control study with the treatment duration of 90 days. Subjects will be recruited into the study based upon the inclusion and exclusion criteria provided. Eligible subjects will be examined for baseline evaluation and lens fitting. Up to sixty (60) subjects will wear the test contact lenses for daily wear and up to twenty-eight (28) subjects will wear the control contact lenses. The subjects will attend seven scheduled study visits and will undergo standard ophthalmic evaluation for contact lens care. The subjects will be followed for a period of three months (90 days) following dispensing of the Test and Control Device.

ELIGIBILITY:
Inclusion Criteria:

Prior to being considered eligible to participate in this study, each subject MUST:

* Be at least 18 years of age as of the date of evaluation.
* Have:

  * read the Informed Consent,
  * been given an explanation of the Informed Consent,
  * indicated an understanding of the Informed Consent and
  * signed the Informed Consent Form.
* Be willing and able to adhere to the instructions set forth in this protocol and able to keep all specified appointments.
* Be a current contact lens wearer.
* Possess wearable and visually functional eyeglasses.
* Be in good general health, based on his/her knowledge.
* Require spectacle lens powers between +10.00 and -10.00 diopters sphere with no more than 2.5 diopters of spectacle refractive astigmatism and be willing to wear lenses in both eyes.
* Have manifest refraction visual acuity equal to or better than 0.10 log MAR (20/25 Snellen) in each eye.

Exclusion Criteria:

Subjects may not be enrolled into the study if ANY of the following apply:

* Subject is wearing lenses in a mono-vision modality and is unwilling to be fit with distance lenses in both eyes. NOTE: Subjects may NOT wear mono-vision lenses at any time during the study as it will interfere with the distance visual acuity measurement.
* Subject appears to exhibit poor personal hygiene (that in the investigator's opinion might prevent safe contact lens wear).
* Subject is currently or within 30 days prior to this study has been an active participant in another clinical study.
* Subject is currently pregnant (to the best of the subject's knowledge), is planning a pregnancy within the next 3 months or is lactating.
* Subject is a member, relative or household member of the office staff, including the investigator(s).
* Subject has a known sensitivity to ingredients used in contact lens care products or over-the-counter lubricants and artificial tears.
* Subject has undergone refractive surgery or is currently receiving or has previously received orthokeratology treatment.
* Subject is aphakic or pseudophakic.
* Subject has ocular or systemic disease such as, but not limited to: anterior uveitis or iritis (past or present), glaucoma, Sjögren's syndrome lupus erythematosus, scleroderma, keratoconus or type II diabetes.
* Subject has 2.5 diopters or great of corneal astigmatism.
* Use of ocular medications for any reason or systemic medications which might interfere with contact lens wear.
* A known history of corneal hypoesthesia (reduced corneal sensitivity).
* Slit lamp findings that would contraindicate contact lens wear, including but not limited to:

  * History of corneal ulcer, corneal infiltrates or fungal infections
  * Corneal scars within the visual axis
  * Pterygium
  * Dry eye symptoms with decrease tear levels and punctate staining ≥ Grade 2
  * Neovascularization or ghost vessels ≥l.5 mm in from the limbus
  * Seborrhoeic eczema, seborrhoeic conjunctivitis
  * History of papillary conjunctivitis that has interfered with lens wear or a current condition of Grade 2 (Mild) or greater
* Clinically significant (Grade 3 or 4) anterior segment abnormalities or any infection of the eye, lids, or associated structures.
* The investigator for any reason considers that it is not in the best interest of the subject to participate in the study.

To be eligible to be randomized for study product trial a subject must have ALL of the inclusion criteria and NONE of the exclusion criteria present. To be eligible for lens dispensing, the subject's study device contact lens visual acuity must be equal to or better than 0.20 log MAR (20/32 Snellen) in each eye

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2020-03-19 (Actual); Study Completion 2020-03-19 (Actual)

PRIMARY OUTCOMES:
Visual Acuity | 90 days
  Comparison of the corrected visual acuity (logMAR) between the Test and Control lens. The working hypothesis is that the visual acuity results will be substantially equivalent between the Test and the Control lenses.
Slit Lamp Exam Observations | 90 days
  Comparison of slit lamp exam findings (scored from 0-4) between Test and Control arms. The working hypothesis is that the findings will be substantially equivalent between the Test and the Control lenses.
Adverse Events | 90 days
  Comparison of the number of device related adverse events in the Test and Control arms. The working hypothesis is that the number of adverse events will be substantially equivalent between the Test and the Control lenses.

SECONDARY OUTCOMES:
Subjective Symptoms | 90 days
  Comparison of subjective symptoms (scored from 0-5) between Test and Control arms. The working hypothesis is that the symptoms will be substantially equivalent between the Test and the Control lenses.

CONTACTS AND LOCATIONS:
Overall Officials: James A Bonafini, BS,MS, Study Chair — Acuity Polymers
Locations (3):
- United States (3):
  - Ala Mona Advanced Eye Clinic, Honolulu, Hawaii
  - Cornea and Contact Lens Institute of Minnesota, Edina, Minnesota
  - Reed Eye Associates, Pittsford, New York